CLINICAL TRIAL: NCT05608187
Title: A Randomized, Double-Blind, Placebo-controlled, Parallel, Exploratory Phase 2a Study to Evaluate Safety and Biological Effect on Wound Healing of ILP100-Topical in Subjects With Diabetic Foot Ulcers
Brief Title: Evaluating Safety and Biological Effect on Wound Healing of ILP100-Topical in Subjects With Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient recruitment issues
Sponsor: Ilya Pharma (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IP-CT-003; 2021-000563-69 (EudraCT Number)
Record Dates: First submitted 2022-10-03; First posted 2022-11-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Wound Heal; Wound Healing Disturbance of; Wound Healing Disorder; Wound Healing Delayed; Diabetic Foot Ulcer; Diabetic Foot Ulcer Mixed
Keywords: emilimogene sigulactibac; ILP100; ILP100-Topical; Lactobacillus reuteri; Limosilactobacillus reuteri; CXCL12; diabetic foot ulcer; wound healing; Ilya Pharma; live biopharmaceutical product; lactic acid bacteria
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, and the allocation of treatments will not be disclosed to subjects, Investigator or Independent Evaluators until database lock after all subjects (who were not withdrawn) completed Week 26.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ILP100Lo (Experimental): During the Treatment Phase, subjects will continue on standard of care according to the protocol and ILP100Lo (ILP100-Topical, 5x10^7 colony forming units (CFU)/cm^2) will be topically administered at two occasions on Day 1 (Baseline and Hour 2), Days 2, 3, and thereafter every second to third day until Day 31.
  Interventions: Biological: ILP100-Topical (emilimogene sigulactibac) 5x10^7 CFU/cm^2
- ILP100Hi (Experimental): During the Treatment Phase, subjects will continue on standard of care according to the protocol and ILP100Hi (ILP100-Topical, 1x10^9 CFU/cm^2) will be topically administered at two occasions on Day 1 (Baseline and Hour 2), Days 2, 3, and thereafter every second to third day until Day 31.
  Interventions: Biological: ILP100-Topical (emilimogene sigulactibac) 1x10^9 CFU/cm^2
- Placebo (Placebo Comparator): During the Treatment Phase, subjects will continue on standard of care according to the protocol and Placebo (ILP100 dilution buffer mixed with the activation peptide SppIP) will be topically administered at two occasions on Day 1 (Baseline and Hour 2), Days 2, 3, and thereafter every second to third day until Day 31.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ILP100-Topical (emilimogene sigulactibac) 5x10^7 CFU/cm^2 — Topical application of ILP100-Topical (emilimogene sigulactibac) at a dose of 5x10^7 CFU/cm^2 wound area.
  Other Names: ILP100-Topical
  Arms: ILP100Lo
Biological: ILP100-Topical (emilimogene sigulactibac) 1x10^9 CFU/cm^2 — Topical application of ILP100-Topical (emilimogene sigulactibac) at a dose of 1x10^9 CFU/cm^2 wound area.
  Other Names: ILP100-Topical
  Arms: ILP100Hi
Biological: Placebo — Topical application of placebo (ILP100 dilution buffer mixed with the activation peptide SppIP).
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel, exploratory phase 2a study to evaluate safety and biologic efficacy on wound healing of ILP100-Topical in subjects with diabetic foot ulcers during 26 weeks with a 5-year long-term follow-up period. A total of 30 subjects will be randomized to low dose of ILP100-Topical (ILP100Lo), high dose of ILP100-Topical (ILP100Hi) or Placebo according to a 1:1:1 randomization schedule.

The study will consist of a 3-weeks Screening and Run-in Phase, followed by a 5-week Treatment Phase starting from Baseline and an Assessment Phase from Week 5 to Week 26. Thereafter, the subjects will be followed yearly during 5 years in a Long-Term Safety Follow-up Phase.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Males and females aged ≥18 years
* Diagnosis of diabetes mellitus type 1 or 2
* HbA1c ≤ 86 mmol/mol (≤ 10%) at Screening
* Subjects with at least one first time or recurrent full thickness ulcer (at or below the ankle) which fulfils all of the following criteria at Screening and at the time of Baseline:

  1. A non-interdigital wound
  2. Accessible for administration of IMP, wound study assessments and procedures
  3. Persistence of the wound for at least 6 weeks at Baseline
  4. Assessed by the investigator to be of non-venous etiology.
  5. Minimum full skin ulcer without undermining, with no exposed muscle, tendon or bone
  6. A wound area of 1.0 - 5.0 cm^2 after sharp or mechanical debridement at Screening
  7. During the 2-weeks between start of Run-in Phase and Baseline the wound size must not decrease by more than 30% or increase by more than 25%, which correspond to wound areas of 0.7 - 6.3 cm^2, or at Screening expected by the Investigator to have a high probability for wound size changes within this range during this period.
* Toe pressure ≥20 mm Hg
* Expected to comply with the study procedures

Exclusion Criteria:

* Infected index wound with clinical signs of inflammation at Screening or Baseline.
* The index wound determined as heavily exuding defined as requiring more than 1 dressing change per day or requiring use of super absorbent dressing
* Wound duration longer than 2 years
* Active Charcot deformity of the study foot
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2
* Hemoglobin concentration <100 g/L at Baseline
* Planned or ongoing treatment with corticosteroids to an equivalent dose of prednisolone >10 mg per day or other immunosuppressive therapy, or such treatment within 4 weeks prior to Baseline
* Has any major surgery or hospitalization planned up to Week 26
* Has changed a treatment for diabetes during the last 3 weeks before Baseline. Dose change is allowed
* Ongoing treatment with dipeptidyl peptidase 4 (DPP-4) inhibitors
* Revascularization procedure in the index wound leg planned or undertaken within 8 weeks before Screening, or under investigation
* Current smokers
* Participation in other clinical studies or having received any investigational treatment within 1 month or at the earliest five times the half-life prior to Screening
* Has any disease conditions, including ulcerative dermatological disorders and vasculitis, or comorbidities which is expected to prevent the subject from participating in the study or confounding the evaluation of the safety profile and effect on wound healing of ILP100
* Pregnant or lactating woman
* Male subjects not willing to use a condom and refrain from donating sperm
* Female subjects of childbearing potential unless they use a contraceptive method with a failure rate of < 1% to prevent pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Compare incidence of adverse events (AEs) between treatment groups | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  The incidence of AEs up to Week 26 will be presented for each treatment group and by category, causality, severity and frequency.
Compare incidence of serious adverse events (SAEs) between treatment groups | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  The incidence of SAEs up to Week 26 will be presented for each treatment group and by category, causality, severity and frequency.

SECONDARY OUTCOMES:
Local tolerability by Investigator's assessment | Compare Investigator's local tolerability assessments up to Week 26 between the ILP100-Topical and Placebo treatment arms.
  Local tolerance to treatment will be assessed by the Investigator. Wound tolerability parameters will be presented in categories of appearance of inflammation, amount of exudate present, hemorrhage, presence of slough/necrotic tissue, presence of granulation tissue and hypergranulation.
Local tolerability by Independent Assessor's assessment | Compare local tolerability up to Week 26 between the ILP100-Topical and Placebo treatment arms.
  Local tolerance to treatment will be assessed by the Independent Assessor. Wound tolerability parameters will be presented in categories of appearance of inflammation, amount of exudate present, hemorrhage, presence of slough/necrotic tissue, presence of granulation tissue and hypergranulation.
Proportion of subjects with a local tolerability parameter Grade ≥ 2 per Investigator's Assessment | Compare the ILP100-Topical and Placebo treatment arms up to Week 26.
  The proportion of subjects with a local tolerability parameter grade ≥ 2 will be calculated (grading system=0 to 3, where 3 is severe). Local tolerance to treatment, infection and wound healing will be assessed by the Investigator. Wound tolerability parameters include appearance of inflammation, amount of exudate present, hemorrhage, presence of slough/necrotic tissue, presence of granulation tissue and hypergranulation.
Proportion of subjects with a local tolerability parameter Grade ≥ 2 per Independent Assessor's Assessment | Compare the ILP100-Topical and Placebo treatment arms up to Week 26.
  The proportion of subjects with a local tolerability parameter grade ≥ 2 will be calculated (grading system=0 to 3, where 3 is severe). Local tolerance to treatment, infection and wound healing will be assessed by the Independent Assessor. Wound tolerability parameters include appearance of inflammation, amount of exudate present, hemorrhage, presence of slough/necrotic tissue, presence of granulation tissue and hypergranulation.
Wound area reduction (percent of Baseline) | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  Wound area will be measured and calculated as proportion of the wound area at Baseline. Metric analyses of wound area is made on 3D models acquired up to Week 26.
Wound healing rate | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  Wound healing rate will be calculated as change in the wound area per week. Wound healing will be assessed by Investigators and Independent Assessor.
Proportion of subjects with ≥50% and 75% partially healed wounds | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  The proportion of subjects with ≥50% and 75% partially healed wounds will be calculated.
Time to partial (≥50% and 75%) and complete healing | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  Time to event outcomes will be evaluated using Kaplan-Meier curves. Wound healing is defined as full skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart. Wound healing will be assessed by Investigators and Independent Assessor.
Wound area | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  Wound area will be measured and calculated (cm^2). Metric analyses of wound healing, including area, are made using 3D models acquired Screening to Week 26. Wound measures will be automatically generated by a computer software and validated by the Independent Assessor.
Proportion of subjects with completely healed wounds | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  The proportion of subjects with completely healed wounds will be calculated. Wound healing is defined as full skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart. Wound healing will be assessed by Investigators and the Independent Assessor.
Proportion of subjects with recurrence of index wound | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  The proportion of subjects with recurrence of index wound will be calculated. For wound assessments after each index wound healing visit, it will be documented if the index wound is still healed or if any recurrence of the wound has occurred.
Proportion of subjects with new wound infections | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  The proportion of subjects with new wound infections will be calculated based on the Investigators evaluation of the skin, including assessing whether there are any new wound infections, at each study visit.
Days on antibiotic treatment | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  Days on antibiotic treatment as a percentage of days in the study up to Week 26 will be calculated for each subject.
Change in subject-reported wound-related pain | Compare ILP100-Topical and Placebo treatment arms up to Week 26
  Change in wound-related pain in the area of the index wound, as reported by subjects, using a numeric rating scale (NRS; 0-10, where 10 is the worst possible pain).
Long-term incidence of AEs. | Compare the ILP100-Topical and Placebo treatment arms up to Year 5 after initiation of treatment.
  AEs and SAEs will be recorded during annual visits from Year 1 through Year 5.
CXCL12 levels in plasma | Compare up to Week 16 between the ILP100-Topical and Placebo treatment arms.
  CXCL12 levels in plasma as measured by enzyme-linked immunosorbent assay (ELISA).
Presence of viable L. reuteri containing the pSIP_CXCL12 plasmid in wounds | Compare up to Year 5 between the ILP100-Topical and Placebo treatment arms.
  Bacteria will be collected from the wound and perilesional skin with sterile cotton swabs which will be cultured.

OTHER OUTCOMES:
Proportion of subjects with index limb amputation and any limb amputation | Compare at Week 26, and thereafter annually Year 1 to 5, between the ILP100-Topical and Placebo treatment arms.
  The proportion of subjects with index limb amputation and any limb amputation will be calculated.
All-cause mortality and index wound-related mortality | Compare at Week 26, and thereafter annually Year 1 to 5, between the ILP100-Topical and Placebo treatment arms.
  Mortality data will be acquired from the patient's medical records.
Quality of life assessed with Wound-Quality of Life (Wound QoL) questionnaire | Compare up to Week 16 between the ILP100-Topical and Placebo treatment arms.
  Quality of life will be assessed by the subjects using the Wound-QoL questionnaire including 17 questions on impairment related to the wound, each to be answered by grades from 0-4 (0='not at all' to 4='very much')
Time for IMP preparation | Compare at Week 4 between the ILP100-Topical and Placebo treatment arms.
  Time needed for IMP preparation, by the study personnel, will be recorded.
Total number of redressings, off-loading and devices used for the treatment of the index wound | Compare the ILP100-Topical and Placebo treatment arms during 16 weeks from baseline.
  Wound management will include redressing, which will be done both during home visits and study site visits, while debridement and changes of off-loading devices should only be done at study site visits. The total number of redressings, off-loading and devices used for the treatment of the index wound will be recorded.
Wound volume | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  Metric analyses of wound healing, including volume, are made using 3D models acquired from Screening to Week 26. Wound measures will be automatically generated by a computer software and validated by the Independent Assessor.
Wound depth | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  Metric analyses of wound healing, including depth, are made using 3D models acquired from Screening to Week 26. Wound measures will be automatically generated by a computer software and validated by the Independent Assessor.
Wound volume reduction (percent of Baseline) | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  Reduction of wound volume (percent of Baseline) will be calculated. Metric analyses of wound healing, including volume, are made using 3D models acquired from Screening to Week 26. Wound measures will be automatically generated by a computer software and validated by the Independent Assessor.
Wound depth reduction (percent of Baseline) | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  Reduction of wound depth (percent of Baseline) will be calculated. Metric analyses of wound healing, including depth, are made using 3D models acquired from Screening to Week 26. Wound measures will be automatically generated by a computer software and validated by the Independent Assessor.
Analyses of predictive factors for wound healing outcome | Analyses of associations between baseline clinical and biologic characteristics and wound healing outcomes up to Week 26.
  Analyses of associations between baseline clinical (including toe pressure at Baseline and sex) and biologic characteristics (including wound size and pH) with wound healing outcomes through Week 26. A statistical regression model will be developed to predict wound healing up to Week 26
Analyses of predictive factors for occurence of AEs | Analyses of associations between baseline clinical and biologic characteristics and occurence of AEs up to Week 26.
  Analyses of associations between baseline clinical (including toe pressure at Baseline and sex) and biologic characteristics (including wound size and pH) with AEs. A statistical regression model will be developed to predict the AE outcome up to Week 26
Analyses of scar area | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  Scar area will be measured for the index wound using 3D models generated from superimposing 2D images and infrared scanning of the topography of the wound and perilesional skin acquired at the study visits.
Analyses of scar volume | Compare between the ILP100-Topical and Placebo treatment arms up to Week 26.
  Scar volume will be measured for the index wound using 3D models generated from superimposing 2D images and infrared scanning of the topography of the wound and perilesional skin acquired at the study visits.
Change from Baseline in level of wound pH | Compare at Weeks 1, 4, 5, 8 and 16 between the ILP100-Topical and Placebo treatment arms.
  Change from Baseline in level of wound pH will be measured on exuding wounds (at the discretion of the Investigator) at selected timepoints just prior to IMP administration using sterile litmus paper strips.
Change from Baseline in local blood flow in wound area measured with Laser Speckle Contrast Analysis | Compare ILP100-Topical and Placebo treatment arms up to Week 16
  Change from Baseline in local blood flow around the index wound will be addressed by non-invasive imaging using Laser Speckle Contrast Analysis (LASCA) where each wound and surrounding skin will be recorded for at least one minute of stable recording at selected timepoints in the study.
Pathogenic wound bacteria characterization upon clinically defined or suspicions of wound infection | Compare species of infection-causing wound pathogens up to Week 26 between the ILP100-Topical and Placebo treatment arms.
  Characteristics of ILP100 will be addressed by collecting bacteria from the wound with sterile cotton swabs which will be cultured.
Wound microbiome profile, including presence and proportion of wound pathogenic bacteria | Compare the microbiome profile up to Week 16 between the ILP100 and Placebo treatment arms.
  The impact of ILP100 on the wound microbiome composition will be assessed from wounds swabs identified by sequencing bacterial 16S ribosomal ribonucleic acid (rRNA) genes.
Presence of anti-drug antibodies (ADA) to CXCL12 and the activation peptide SppIP up to Year 5 | Compare presence of ADA up to Year 5 between the ILP100-Topical and Placebo treatment arms.
  The development of anti-drug antibodies (ADAs, to CXCL12 and SppIP) as measured by electrochemiluminescence immunoassay (ECLIA).
Analysis of L. reuteri containing the pSIP_CXCL12 plasmid in blood, feces, and perilesional skin | Analyses of presence of L. reuteri containing the pSIP_CXCL12 plasmid up to Year 5.
  Shedding to the external environment will be measured in feces and water lock samples collected at the sites. The method will determine the number of live L. reuteri R2LC containing pSIP_CXCL12 in the samples. Used dressings will also be collected for shedding analyses of L. reuteri R2LC containing the pSIP_CXCL12 plasmid.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Apelqvist, MD/PhD, Principal Investigator — Department of Endocrinology, Skåne University Hospital, Malmö, Sweden
Locations (2):
- Sweden (2):
  - Department of Endocrinology, Skåne University Hospital, Lund
  - Clinical Diabetes Research Unit at Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided
Undecided due to ongoing development.

REFERENCES:
- [Background] Vagesjo E, Ohnstedt E, Mortier A, Lofton H, Huss F, Proost P, Roos S, Phillipson M. Accelerated wound healing in mice by on-site production and delivery of CXCL12 by transformed lactic acid bacteria. Proc Natl Acad Sci U S A. 2018 Feb 20;115(8):1895-1900. doi: 10.1073/pnas.1716580115. Epub 2018 Feb 5. PMID 29432190
- [Background] Ohnstedt E, Lofton Tomenius H, Vagesjo E, Phillipson M. The discovery and development of topical medicines for wound healing. Expert Opin Drug Discov. 2019 May;14(5):485-497. doi: 10.1080/17460441.2019.1588879. Epub 2019 Mar 14. PMID 30870037
- [Background] Ohnstedt E, Lofton Tomenius H, Frank P, Roos S, Vagesjo E, Phillipson M. Accelerated Wound Healing in Minipigs by On-Site Production and Delivery of CXCL12 by Transformed Lactic Acid Bacteria. Pharmaceutics. 2022 Jan 19;14(2):229. doi: 10.3390/pharmaceutics14020229. PMID 35213962